CLINICAL TRIAL: NCT05943964
Title: A Pilot Study of Virtual Rehabilitation After Hematopoietic Cell Transplantation
Brief Title: Virtual Rehabilitation in HCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Muna Qayed, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005995
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic Cell Transplant
Keywords: Virtual Rehabilitation; Virtual Exercise; Physical fitness
MeSH Terms: interventions — Rehabilitation; Telerehabilitation; Hematocrit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual exercise and rehabilitation program (Experimental): Trial of exercise and rehabilitation program delivered via a virtual platform for patients undergoing HCT at Children's Healthcare of Atlanta.
  Interventions: Behavioral: Virtual exercise and rehabilitation program

INTERVENTIONS:
Behavioral: Virtual exercise and rehabilitation program — Participants will have two 30-minute sessions per week for 12 weeks. The program will focus on aerobic exercises and stretching exercises. When applicable, stretching exercises will focus on areas of contractures, and joints with limited range of motion (ROM).
  Sessions will be completed by a team of Physical Therapists using the established telemedicine platform at Children's Healthcare of Atlanta, as used routinely in the blood and marrow transplant clinic for clinical care (Epic). Adherence to the program will be encouraged during monthly standard clinic visits.
  Other Names: Virtual Rehabilitation in HCT

SUMMARY:
Chronic GVHD (cGVHD) is a major cause of illness in patients who undergo hematopoietic transplantation (HCT). GVHD can affect any organ in the body, can require several years of treatment, and can impact the quality of life (QoL). Physical activity and exercise have been shown to enhance fitness and improve QoL in chronic illnesses including GVHD, however, patients often have barriers to attending sessions including distance, risk of infection, and physical therapists' lack of experience with pediatric patients. The team's goal is to assess whether a virtual rehabilitation program in children post-HCT (including children with chronic GVHD) is feasible and whether its implementation will improve physical functioning and QoL. Patients between the ages of 8 and 23 years who are at least one hundred days post-HCT will be eligible for participation. Patients will have an assessment by a pediatric physical therapist at the time of study entry, at the end of the rehabilitation program, and approximately 3 months later. They will be supplied with some exercise equipment (such as dumbbells and resistance bands). Patients will have twice weekly half-hour one-on-one online sessions with the physical therapist for 12 weeks. Patients will be recruited through the bone marrow transplant clinic.

DETAILED DESCRIPTION:
Physical rehabilitation is an important, but often inadequately addressed, component of comprehensive cGVHD care. Physical activity and exercise have been shown to enhance fitness and improve QoL, including in patients with chronic diseases. Studies in patients undergoing HCT (including patients with GVHD) show the positive impact of exercise on QoL including improved endurance, muscular strength, functional capacity, perceptions of fatigue, and emotional, and social well-being. Evidence supports that the most effective intervention is supervised participation, followed by self-administered exercise programs and that these interventions are safe and well-tolerated. While rehabilitation is often specifically recommended to cGVHD patients, barriers include the ability to travel, and the time and distance from the rehabilitation center. This is especially relevant in pediatrics, where fewer centers offer services to children. Additionally, parents and providers often express concerns about infection risk as a strong barrier to pursuing rehabilitation. The use of a virtual platform overcomes these limitations.

Virtual cardiac rehabilitation programs are a novel concept designed to improve accessibility and adherence. These have been shown to be beneficial in some studies post-cardiac transplantation. Investigators propose a virtual program that incorporates exercise and stretching for children with cGVHD. If successful, this could be a guide for institutions to adopt and could help improve the landscape of rehabilitation in pediatric and adult patients with cGVHD. Further, patients early post-HCT often benefit from rehabilitation services, however, these services are often limited by the extensive outpatient visit schedule, acute illness, and concern regarding isolation and severely immunocompromised state. If feasible, this virtual program could be extended to patients post-HCT without cGVHD and is likely to improve daily function and QoL.

ELIGIBILITY:
Inclusion Criteria:

* Recipients between the ages of 8 and 23 years ≥100 days post allogeneic HCT.
* Patients 8-14 years old should have a caregiver willing to assist with the implementation of the exercises during the session
* Patients should have access to devices and a reliable internet connection.
* Patients should be cleared for exercise by their physician
* Patients are eligible to participate regardless of underlying diagnosis, preparative regimen, or graft source.

Exclusion Criteria:

* Any physical impediment to exercise as evaluated by the treating physician.
* Non-English-speaking patients (due to a lack of available interpreters through the telemedicine platform).

Ages: 8 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adherence Rate | Throughout the intervention (up to 16 weeks)
  Percentage of sessions completed per participant. A log will be kept to track the sessions completed by participants during the study participation
Feasibility of the rehabilitation program | Up to 4 years
  Percentage of patients completing ≥75% of sessions

SECONDARY OUTCOMES:
Change in 6-minute walk test at completion of the rehabilitation program | Baseline and up to 16 weeks
  The 6-Minute Walk Distance (6MWD) test measures the distance, in meters, that a patient can quickly walk on a flat, hard surface in a period of 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Muna Qayed, MD, MsCR, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No